CLINICAL TRIAL: NCT02275273
Title: Adnexal Masses : Correlation Between MRI (Magnetic Resonance Imagery) and Anatomopathology
Status: Completed | Type: Observational
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Carine DE PREZ, PMD, Brugmann University Hospital
Other Study IDs: Adnexal masses
Record Dates: First submitted 2014-06-27; First posted 2014-10-27 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Adnexal Masses
Keywords: Adnexal Masses; Magnetic Resonance Imaging; Anatomopathology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with adnexal masses: Every patient that are at least 18 years old with a planned pelvic magnetic resonance imagery and an adnexectomy within the institution.

SUMMARY:
The goal of this study is to correlate the pelvic magnetic resonance imagery characteristics of adnexal masses with their anatomopathological characteristics.

DETAILED DESCRIPTION:
Several studies have identified the characteristics of adnexal masses obtained by different imaging techniques (echography, scanner and magnetic resonance) and corresponding to benign, borderline or malign masses (Kurtz et al 1999, Grabowska-Derlatka et al, 2013, Tanaka et al 2011, Asch et al 2008).

Recently, studies have even established ecographic and magnetic resonance imaging scores combining these characteristics (Thomassin-Naggara 2013, Timmerman 2005), some of these characteristics being considered as more suspect than others.

However, these studies have considered adnexal masses in their globality only and to our knowledge, none have correlated their imagery characteristics with their precise anatomopathology characteristics.

The goal of this study is thus to correlate the pelvic magnetic resonance imagery characteristics of the adnexal masses with their anatomopathology characteristics, in order to add complementary information for the future management of masses that are defined as borderline according to imagery.

ELIGIBILITY:
Inclusion Criteria:

- Every woman aged 18 years and more, with a planned pelvic magnetic resonance imagery and a planned adnexectomy within the institution.

Exclusion Criteria:

- Insufficient technical quality of the pelvic magnetic resonance imagery images or of the anatomopathological analysis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with adnexal masses, with a planned pelvic magnetic resonance imagery and a planned adnexectomy within the institution, having signed the informed consent form.
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2014-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
RECIST criteria | at MRI diagnosis
  MRI imaging (standard protocol for ovarian pathology). The MRI will be realised on a 3.0T instrument (Philips Medical Systems, Best, The Netherlands). The patient will be placed in dorsal decubitus with an antenna placed at the pelvic level. Just before the examination, Buscopan IV will be injected. The initial protocol will consist in a localisation examination followed by a standard protocol for ovarian pathologies, meaning a SE T2WI in the three plans, an axial diffusion sequence and a pondered T1 sequence (T1 dynamic contrast imaging). The total examination time will be 20 minutes on average.
Percentage of epithelial and conjunctive zones in the adnexal mass obtained by surgery | 24h after MRI diagnosis
  The anatomopathologist will contact the surgeons when an adnexectomy is programmed. A detailed macroscopic description is realized (photographies of the external capsule) and the fragment is oriented according to 6 axes (superior, inferior, external, internal, anterior, posterior) with permanent tissues marking dyes. The piece will be sectioned in 1cm slices, a picture of each one being taken. The piece will be fixed in formol and embedded in paraffin. Slices will be made using a RM 2235 Leica Microtome and colored with hematoxylin/eosin, for examination by the anatomopathologist. The radiologist and the anatomopathologist will select, by consensus, interest zones that will be examined with an accredited microscope (ISO9001 accreditation). Several parameters such as the percentage of epithelial and conjunctive zones will be observed, described and semi-quantified. Immunomarkings will be realized if necessary, according to the criteria described in the ISO9001 accreditation files.

CONTACTS AND LOCATIONS:
Overall Officials: Carine De Prez, Chef de service, Study Director — CHU Brugmann; Françoise HULET, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

REFERENCES:
- [Background] Kurtz AB, Tsimikas JV, Tempany CM, Hamper UM, Arger PH, Bree RL, Wechsler RJ, Francis IR, Kuhlman JE, Siegelman ES, Mitchell DG, Silverman SG, Brown DL, Sheth S, Coleman BG, Ellis JH, Kurman RJ, Caudry DJ, McNeil BJ. Diagnosis and staging of ovarian cancer: comparative values of Doppler and conventional US, CT, and MR imaging correlated with surgery and histopathologic analysis--report of the Radiology Diagnostic Oncology Group. Radiology. 1999 Jul;212(1):19-27. doi: 10.1148/radiology.212.1.r99jl3619. PMID 10405715
- [Background] Grabowska-Derlatka L, Derlatka P, Palczewski P, Danska-Bidzinska A, Pacho R. Differentiation of ovarian cancers from borderline ovarian tumors on the basis of evaluation of tumor vascularity in multi-row detector computed tomography--comparison with histopathology. Int J Gynecol Cancer. 2013 Nov;23(9):1597-602. doi: 10.1097/IGC.0b013e3182a80a41. PMID 24172096
- [Background] Tanaka YO, Okada S, Satoh T, Matsumoto K, Saida T, Oki A, Yoshikawa H, Minami M. Solid non-invasive ovarian masses on MR: histopathology and a diagnostic approach. Eur J Radiol. 2011 Nov;80(2):e91-7. doi: 10.1016/j.ejrad.2010.05.032. Epub 2010 Jun 23. PMID 20576386
- [Background] Asch E, Levine D, Kim Y, Hecht JL. Histologic, surgical, and imaging correlations of adnexal masses. J Ultrasound Med. 2008 Mar;27(3):327-42. doi: 10.7863/jum.2008.27.3.327. PMID 18314510
- [Background] Thomassin-Naggara I, Aubert E, Rockall A, Jalaguier-Coudray A, Rouzier R, Darai E, Bazot M. Adnexal masses: development and preliminary validation of an MR imaging scoring system. Radiology. 2013 May;267(2):432-43. doi: 10.1148/radiol.13121161. Epub 2013 Mar 6. PMID 23468574
- [Background] Timmerman D, Testa AC, Bourne T, Ferrazzi E, Ameye L, Konstantinovic ML, Van Calster B, Collins WP, Vergote I, Van Huffel S, Valentin L; International Ovarian Tumor Analysis Group. Logistic regression model to distinguish between the benign and malignant adnexal mass before surgery: a multicenter study by the International Ovarian Tumor Analysis Group. J Clin Oncol. 2005 Dec 1;23(34):8794-801. doi: 10.1200/JCO.2005.01.7632. PMID 16314639